CLINICAL TRIAL: NCT02093871
Title: A Phase 1 Trial of Perfusion Induced Systemic Hyperthermia (PISH) Over Multiple Cycles for Terminal Ovarian Cancer
Acronym: PISH-2
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: ThermalCore Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thermalcore-01
Record Dates: First submitted 2013-08-14; First posted 2014-03-21 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Therapeutic hyperthermia; HEATT; whole body hyperthermia; hyperthermia; PISH; Verthermia; Phase 1 clinical trial; stage 3 ovarian cancer; stage 4 ovarian cancer; stage III ovarian cancer; stage IV ovarian cancer; late stage ovarian cancer; Core HFC; Lilja; Vertrees; Bastidas; total body hyperthermia
MeSH Terms: conditions — Ovarian Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ThermalCore Hyperthermia System (Experimental): Patients will undergo 6 cycles of therapeutic hyperthermia with the ThermalCore Perfusion Induced Systemic Hyperthermia System every 28 days
  Interventions: Device: ThermalCore Hyperthermia System

INTERVENTIONS:
Device: ThermalCore Hyperthermia System — Patients will undergo 6 cycles of therapeutic hyperthermia with the ThermalCore Perfusion Induced Systemic Hyperthermia System every 28 days

SUMMARY:
To confirm the safety of 6 cycles of Perfusion Induced Systemic Hyperthermia (PISH) provided every 28 days in 3rd line ovarian cancer patients.

DETAILED DESCRIPTION:
This study is a prospective, single-arm phase I trial of 20 ovarian cancer patients to be treated with PISH for 6 cycles, delivered every 28 days. This mimics chemotherapy treatments, in concordance with the fractional cell kill hypothesis of cytotoxic agents.

As this study is for safety, only, metastatic peritoneal or ovarian cancer, of any histology (epithelial, sex-cord stromal, germ cell, or sarcoma) that has progressed after 2 cycles of chemotherapy, and is considered incurable, will be included. All patients must meet performance status and organ function entry criteria. Patients must have first undergone standard first line primary surgery and chemotherapy, and have then gone on to fail second line chemotherapy treatment, (with or without secondary cytoreductive surgeries). Patients must be candidates for, and expecting treatment by, the usual third line chemotherapy agent palliation traditionally offered by medical oncology. Patients may have received treatment beyond third-line therapy, as long as they meet entry requirements for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with ovarian cancer/primary peritoneal cancer of any histologic subtype, including epithelial, germ cell, sex-cord stromal, or sarcoma.
* Failure of first line surgery and chemotherapy, AND at least second line chemotherapy, with or without secondary cytoreductive surgeries
* Patients must be eligible for, and be expecting treatment by, an FDA approved chemotherapy regimen commonly used for their disease as per community standard.
* Female patients, aged 18-69 years old, and must be aware of the investigational nature of this treatment, and then indicate informed consent by the IRB-approved written process.
* All patients must have a performance status (Karnofsky score) greater than 80
* Patients may have been treated with radiotherapy, or non-chemotherapy anti-neoplastics (e.g. anti-angiogenic agents like bevicizumab)
* Hematologic Parameters: WBC of > 4,000/μl with an ANC >1500/μl, and a Platelet count of >100,000/μl
* Renal Filtration: pretreatment measured or calculated creatinine clearance of > 50 ml/minute by Cockroft-Gault equation or MDRD
* Electrolytes parameters: Patients pre-treatment serum calcium be in the normal (8.5-10.5 mg/dL) range.
* Liver function parameters: Bilirubin ≤ 1.5 times upper limit of normal (ULN); AST and ALT ≤ 2.5 times ULN; Alkaline phosphatase ≤ 2.5 times ULN; PT/INR ≤ 1.5 times ULN (or an in-range INR, usually between 2 and 3, if the patient is on a stable dose of therapeutic warfarin)

Exclusion Criteria:

* Patients who would be expected to receive benefit, on third recurrence, by a platinum-based regimen of chemotherapy
* Uncontrolled hypertension, defined as systolic BP > 160 mm Hg or diastolic BP > 100 mm Hg
* Myocardial infarction or unstable angina within the past 6 months
* NYHA class II-IV congestive heart failure
* Atrial fibrillation (AF) or Supra Ventricular Tachycardia (SVT) whether controlled by drugs or not; Any other serious arrhythmia, requiring medication to control
* Currently on anticoagulation for DVT or PE.
* Peripheral vascular disease ≥ CTCAE grade 2 (at least brief [< 24 hrs] episodes of ischemia managed non-surgically and without permanent deficit)
* CNS metastases
* Lung disease, and a pulmonary function test (PFT) with FEV1 <50% expected.
* Patients who have been treated with any chemotherapy or biologic therapy within the previous 21 days.
* Subjects who are unable or unwilling to comply with the follow-up schedule and requirements or sign informed consent

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Organ toxicity | 28 days
  Patients continue to meet the entry criteria for organ toxicity defined in the trial by the time prior to next scheduled treatment at 28 days.

SECONDARY OUTCOMES:
Time To Progression of Disease | 8 months
  Time To Progression (TTP, defined as the interval from treatment initiation to disease progression) for the cohort. Measurement of Time To Progression (TTP) for the cohort will be conducted using PET CT, CA-125, and physical examination. Progression is defined as radiologic progression RECIST criteria, CA-125 doubling per Gynecologic Intergroup Definition of progression of disease, or any evidence of palpable lesion growth on physical examination.

OTHER OUTCOMES:
Number of patients with unexpected serious adverse events | 8 Months
  Determine the frequency and severity of unexpected serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jan Winetz, MD, Principal Investigator — ThermalCore Inc
Locations (1):
- Good Samaritan Hospital, San Jose, California, United States